CLINICAL TRIAL: NCT04854304
Title: Supplemental Screening for Breast Cancer With Abbreviated Breast MR for Black Women With Increased Breast Density
Brief Title: Abbreviate or FAST Breast MRI for Supplemental Breast Cancer Screening for Black Women at Average Risk and Dense Breasts
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 844978
Record Dates: First submitted 2021-04-08; First posted 2021-04-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Diseases
Keywords: Black women; dense breast
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fast Breast Abbreviated Magnetic Renounce Imaging — Fast Breast MRI Imaging

SUMMARY:
500 patients will be prospectively recruited to undergo a fast breast MRI examination. The women will be recruited for the study will meet the following criteria: 1. African American 2. negative DBT examination 11 months prior to recruitment 3. Heterogeneously and Extremely breast densities 4. clinically asymptomatic- no palpable masses, focal thickening or clinically significant discharge. Investigators will identify these patients EPIC database utilizing the date of their last mammogram. Interested patients may contact our research coordinators by the phone number provided in the recruitment materials. The study recruitment information will also be shared with referring physicians. Physicians may also directly refer patients to the study.

DETAILED DESCRIPTION:
500 patients will be prospectively recruited to undergo an abbreviated or "FAST" breast MRI examination. The women will be recruited for the study must meet the following criteria: 1. African American 2. negative DBT examination no more than 11 months prior to the FAST MR 3. Heterogeneously and Extremely breast densities as graded on their most recent mammogram 4. clinically asymptomatic- no palpable masses, focal thickening or clinically significant nipple discharge. Investigators will identify these women via the EPIC database utilizing the date of their last mammogram. Interested women may contact our research coordinators by the phone number provided in the recruitment materials. The study recruitment information will also be shared with referring physicians. Physicians may also directly refer patients to the study.

ELIGIBILITY:
Inclusion Criteria:

1. African American female
2. Negative DBT examination within eleven months prior to recruitment
3. Heterogeneoulsy and Extremely breast densities
4. Clinically asymptomatic- no palpable masses or focal thickening, etc.

Exclusion Criteria:

1. Patients who are pregnant and lactating
2. Patient who have not had a mammogram (DBT) in the past 11months
3. Patients who are unwilling or unable to provide written informed consent
4. Patients symptomatic for breast disease (e.g. experiencing discharge, lumps, ect.)
5. Recent breast surgery in the past 2 years including breast enhancements (e.g. implants or injections)
6. Patients who are unable to received an MRI with Gadolinium contrast
7. Patients who have not had an MRI of the breast with the past year

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female at birth
Study Population: Women who have no personal history and no family history of Breast Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2027-12-13 (Estimated); Study Completion 2028-07-13 (Estimated)

PRIMARY OUTCOMES:
Breast cancer detection and false negative rates of supplemental screening with AB-MR | Through the completion of study, an average of 4 year
  The cancer detection and false negative rate (per 1000 women screened) of supplemental screening with AB-MR in this population will be measured as well as the stage, grade and subtype of detected and non-detected breast cancers.
Additional screening outcomes | Through the completion of study, an average of 4 year
  The rates of false positive exams prompting biopsy and short term follow-up recommendations after AB-MR will be evaluated.

SECONDARY OUTCOMES:
The screening outcomes of AB-MR in this population of Black women will be compared to a similar population of Caucasian women undergoing AB-MR. | Through the completion of study, an average of 4 year
  The cancer detection, false negative and false positive rates as well as stage and subtypes of cancers will be compared to a similar population of Caucasian women screened with AB-MR

CONTACTS AND LOCATIONS:
Overall Officials: Emily F Conant, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- UPENN, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No